CLINICAL TRIAL: NCT03807583
Title: Prospective, Monocentric, Open-label, Randomized Study Comparing Intradialytic Plasma Kinetics of Amino Acids After Administration Per os of Renoral® and Intravenous Administration of Amino Acids.
Brief Title: Plasma Amino Acid Levels After Protein Ingestion or Amino Acid Injection During Dialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indigo Therapeutics (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ID-RCB 2018-00145-50
Record Dates: First submitted 2018-12-27; First posted 2019-01-17 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: End Stage Renal Disease on Dialysis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: This clinical study is a monocentric, randomized, open-label, 3 parallel arms, and controlled study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention)
- AMINOVEN® 10% (Active Comparator): The AMINOVEN® 10% comparative product is a drug in the form of a 130 mL intravenous infusion solution. This product is composed of amino acids.
  The product is administered per os during the first hour of dialysis sessions for the duration of the study.
  Interventions: Drug: Aminoven 10%
- RENORAL® (Experimental): The product under study RENORAL® is notified to the DGCCRF with the status of food supplement for medical purposes (FSMP) and specific for renal insufficiency.
  The product is a beverage packaged in 150 mL aluminum cans. It contains a liquid solution of native milk proteins and partially hydrolyzed whey proteins.
  Interventions: Dietary Supplement: RENORAL

INTERVENTIONS:
Drug: Aminoven 10% — After randomization to the visit Day 60, two months after patients inclusion (Visit Day 0) and one month after clinical examination (Visit Day 30), patients will be assigned to a group:
  * group A: RENORAL® product
  * group B: AMINOVEN® 10% product
  * group C: control group (without intradialytic supplementation)
  Patients will consume the products and will be followed for 3 months, one visit per month (Day 90, Day 120, Day 150). Protocol visits are included in the patient's course of care.
  Arms: AMINOVEN® 10%
Dietary Supplement: RENORAL — After randomization to the visit Day 60, two months after patients inclusion (Visit Day 0) and one month after clinical examination (Visit Day 30), patients will be assigned to a group:
  * group A: RENORAL® product
  * group B: AMINOVEN® 10% product
  * group C: control group (without intradialytic supplementation)
  Patients will consume the products and will be followed for 3 months, one visit per month ( V3, V4, V5). Protocol visits are included in the patient's course of care.
  Arms: RENORAL®

SUMMARY:
The aim of the study is to compare intradialytic plasma kinetics of amino acids after administration per os of Renoral or intravenous administration of amino acids in patients with end-stage renal disease treated with hemodialysis maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 (limit included),
* Patients treated with hemodialysis for at least 3 months (limit included),
* Patient with normal albuminemia ≥ 35 g/L
* Patient capable and willing to comply with the protocol and willing to give written informed consent,
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* Patient with a known food allergy or intolerance,
* Patient with alcohol consumption ≥ 20 g/day (equivalent to 2 glasses per day),
* Patient following a specific diet (vegetarian, hypocaloric, restrictive gluten-free diet....) outside the high-protein diet of the patient with terminal renal insufficiency or deviant behavior,
* Pregnant or breastfeeding woman or intending to become pregnant within the next 3 months
* Patient taking vitamin or mineral supplementation for less than one month,
* Patient participating in another clinical study or in a period of exclusion from a previous clinical study;
* Patient refusing to give written consent,
* Patient not able to read and understand information, consent or other study related documents (self-administered questionnaires),
* Patient unable to give informed consent,
* Patient deprived of liberty by administrative or judicial decision, under guardianship or curatorship.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Plasma total amino acid concentration | Day 60; Time 240 minutes of the kinetic
  The efficacy of the test product will be evaluated by comparing this criterion between the RENORAL® and AMINOVEN® groups.

SECONDARY OUTCOMES:
Plasma total amino acid concentration | Day 60; Time 240 minutes of kinetics
  Comparison between the RENORAL® group and the plasma total amino acid concentration control group
Plasma total amino acid concentration | Time 0 minutes, Time 60 minutes and Time 120 minutes of kinetics
  Comparison between the RENORAL® group and each AMINOVEN® group and control
Plasma total amino acid concentration | Day 90; Day 120 and Day 150 at time 240 minutes of kinetics
  Comparison between the RENORAL® group and each AMINOVEN® group and control
Protein catabolism | Day 90; Day 120 and Day 150 at time 0 minutes of kinetics
  Plasma urea concentration (mmol.L-1) ;
Protein catabolism | Day 90; Day 120 and Day 150 at time 0 minutes of kinetics
  Plasma creatinine concentration (µmol.L-1);
Protein catabolism | Day 90; Day 120 and Day 150 at time 0 minutes of kinetics
  Standardized protein catabolism rate (nPCR) (g/kg/day):
  * BUN: Blood urea nitrogen is one of the main renal function parameters (mmol/L).
  * ID Refers to the interdialytic period in hours.
  * ID BUN rise refers to the registered change in blood urea nitrogen during the interdialytic period.
  The two nPCR formulas used are:
  nPCR Anuric = 0.22 + (0.864 x (ID BUN rise in mg/dL) / (ID hours)) nPCR Total = nPCR Anuric + (Urine urea nitrogen in g x 150) / (ID hours x Weight in kg)
Inflammation degree | Day 90; Day 120 and Day 150 at time 0 minutes of kinetics
  Comparison between the RENORAL® group and each AMINOVEN® group and control. Evaluated by plasma CRPus concentration (mg.L-1).
Nutritional status | Day 90, Day 120 and Day 150; At time 0 minute of kinetics
  Plasma albumin concentration (g.L-1) ;
Nutritional status | Day 90, Day 120 and Day 150; At time 0 minute of kinetics
  - Plasma prealbumin concentration (g.L-1) ;
Nutritional status | Day 90, Day 120 and Day 150; At time 0 minute of kinetics
  - Plasma ferritin concentration (µg.L-1) ;
Nutritional status | Day 90, Day 120 and Day 150; At time 0 minute of kinetics
  - Plasma transferrin concentration (ng.L-1) ;
Nutritional status | Day 150
  - Body mass index (BMI) (kg/m2)
Nutritional status | Day 150
  - Body composition by impedance measurement (Body Composition Monitor / Fresenius Medical Care) analyzed by the following parameters: lean mass (LTM) (kg), fat mass (ATM) (kg) and water overload (OH) (L)
Nutritional status | During the week preceding Day 150
  - Total energy intake (average of the 3 food survey days, kcal/day);
Nutritional status | During the week preceding Day 150
  - Protein consumption (average of the 3 food survey days, g/day)
Muscular force | Day 150
  Evaluated by the gripping force by dynamometry (kg)
Acceptability of Renoral® | Day 60 and Day 150
  Self-administered questionnaire
  4 questions:
  * Overall, do you like this product? minimum score:1 (I don't like); maximum score: 9 (I like a lot)
  * How do you find the texture of the product? Score 1: Not at all pleasant Score 2: Somewhat unpleasant Score 3: Somewhat pleasant Score 4: Very pleasant
  * What do you think of the practicality of the product? Score 1 - Not practical at all Score 2 - Not very practical Score 3 - Somewhat practical Score 4 - Very practical
  * What do you think of the vanilla flavour of the product? Score 1 - Much too pronounced Score 2 - Somewhat pronounced Score 3 - Just the right way Score 4 - Not strong enough Score 5 - Really not pronounced

OTHER OUTCOMES:
Blood pressure (mmHg) | Day 0 to Day 150 at time 0, 60, 120 and 240 minutes of dialysis
  Security parameters evaluated from Day 0 to Day 150
Blood count | Day 0 to Day 150 at time 0 minute
  Security parameters evaluated at all visits (from Day 0 to Day 150)
Blood sugar | Day 0 to Day 150 at time 0 minute
  Security parameters evaluated at all visits (from V0 to V5)
Electrolyte balance by ionogram. Blood ionogram expressed in (mmol.L-1), the parameters considered are: Sodium, Potassium, Chlorine, Bicarbonates, Calcium, and Phosphorus. | Day 0 to Day 150 at time 0 minute
  Security parameters evaluated at all visits (from V0 to V5)
Liver function (Alkaline Phosphatase concentration) | Day 0 to Day 150 at time 0 minute
  Security parameters evaluated at all visits (from V0 to V5)
Thyroid function (PTH concentration) | Day 0 to Day 150 at time 0 minute
  Security parameters evaluated at all visits (from V0 to V5)

CONTACTS AND LOCATIONS:
Overall Officials: RAYMOND AZAR, MD, Principal Investigator — HOSPITAL CENTER DUNKERQUE
Locations (1):
- Hopital Center, Dunkirk, France

IPD SHARING:
Plan to Share IPD: No